CLINICAL TRIAL: NCT01914523
Title: Comparison of the Macintosh, King Vision®, Glidescope® and AirTraq® Laryngoscopes in Routine Airway Management
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KFHU-FBR 0039
Record Dates: First submitted 2013-07-28; First posted 2013-08-02 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Patients Need Tracheal Intubation
Keywords: Laryngoscope; Macintosh; Glidescope; King Vision; AirTraq; tracheal intubation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Macintosh (Placebo Comparator): tracheal intubation will be performed using a Macintosh
  Interventions: Device: Macintosh
- King Vision (Active Comparator): tracheal intubation will be performed using a King Vision
  Interventions: Device: King Vision
- Glidescope (Active Comparator): tracheal intubation will be performed using a Glidescope
  Interventions: Device: Glidescope
- AirTraq (Active Comparator): tracheal intubation will be performed using a AirTraq
  Interventions: Device: AirTraq

INTERVENTIONS:
Device: Macintosh — Laryngeal exposure and tracheal intubation using that device
  Arms: Macintosh
Device: King Vision — Laryngeal exposure and tracheal intubation using that device
  Arms: King Vision
Device: Glidescope — Laryngeal exposure and tracheal intubation using that device
  Arms: Glidescope
Device: AirTraq — Laryngeal exposure and tracheal intubation using that device
  Arms: AirTraq

SUMMARY:
Failure to successfully intubate the trachea and secure the airway remains a leading cause of morbidity and mortality, in the operative [1-2] and emergency settings. [3-4]. When the concept of endotracheal intubation was developed, 100 years ago the procedure was performed blindly. Shortly thereafter, laryngoscopes were invented, allowing for direct visualization of the larynx with a viewing angle of 15 degrees [5]. Insufficient laryngoscopic view constitutes the main reason for difficult intubations [6].

Video laryngoscopes provide an improved view of the glottis, as the camera is a few millimeters away from the glottis. The use of Glidescope [7-8] and AirTraq [9] laryngoscopes has superior glottis view and ease of tracheal intubation compared with the traditional Macintosh laryngoscope. Unfortunately, the use video laryngoscopes is associated with longer time to tracheal intubation compared with the traditional techniques which be explained with the variable learning curves of the practitioners. [10]

The King Vision video laryngoscope® (King Systems Company, a division of Consort Medical, Indianapolis, Indiana, USA) is a relative newcomer to the video laryngoscopes of devices that claim to provide the "perfect view" for intubation via use of video and digital technology.

The King Vision Video laryngoscope is a two piece design. It has a reusable monitor that attaches to disposable blades. Blades are made of high quality poly-carbonate plastic and house a complementary semi-conductor (CMOS) micro camera offers a 160 degree of view and LED light source.

Up to best of the authors' knowledge, there is no current published or ongoing randomized controlled comparative study of the use of King Vision laryngoscope with traditional laryngoscope and other video laryngoscopes for endotracheal intubation.

DETAILED DESCRIPTION:
Eighty six ASA I-II patients aged 18-65 years scheduled for elective minor surgery under general anesthesia who need tracheal intubation will be included in this prospective, randomized, single-blind, controlled study at the author's center after obtaining approval of the local ethical committee and an informed written consent from all participants.

Patients will be randomly allocated to one of four groups (n=30 for each) namely, Macintosh, King Vision, Glidescope, or AirTraq groups, by drawing sequentially numbered sealed opaque envelopes containing a software-generated randomization code (Random Allocation Software, version 1.0.0, Isfahan University of Medical Sciences, Isfahan, Iran).

Anesthesia:

The Mallampati airway score, thyromental and sternomental distances with neck extension, and the degree of mouth opening will be evaluated preoperatively as factors predicting difficult intubation. Patients' monitoring includes pulse oximetry, noninvasive blood pressure electrocardiography, state and response Entropy (SE and RE) and train of four (TOF) before induction of anesthesia.

The intubators who will participate in the study received a standardized manikin based training course followed by 10 successful intubations in clinical practice with the use of Macintosh, King Vision®, Glidescope®, and the Airtraq® laryngoscopes for endotracheal intubation.

Anesthetic technique will be standardized in all studied. After breathing 100% oxygen for 3 min through a facemask in a supine "sniffing" position, all patients will receive intravenous propofol 2-3 mg/kg and remifentanail 0.05-0.25 µg/kg/min for induction of anesthesia until loss of consciousness defined as decrease of SE less than 50 and the difference between RE and SE is less than 10. Rocrunium 0.6 mg.kg will be administered and complete relaxation will be monitored using a nerve stimulator (TOF-GE, Datex-Ohmeda Division, Instrumentarium Corporation, Helsinki, Finland).

The studied data during intubation will be collected by an independent investigator; the intubator will not informed about the time taken to achieve any intubations. Tracheal intubation will be performed with the Macintosh, King Vision, Glidescope, or AirTraq laryngoscopes, according to the assigned randomization code.

Time to tracheal intubation, defined as the time when the investigated laryngoscope passes the central incisors to the time when the tip of the tracheal tube passed through the glottis, will be determined. The duration of laryngoscopy, defined as the time from holding of the investigated laryngoscope to the appearance of as the first upward deflection on the capnograph, will be recorded.

Before each procedure, the capnograph gas sample delay time will be measured and then subtracted from total recorded duration of laryngoscopy, to correct for the different sampling times between the capnographs used. [11] The best view during laryngoscopy (using Cormack and Lehane classification) will be recorded. [12]

If intubation is unsuccessful at the first attempt, took longer than 120 seconds, or if desaturation noted on the pulse oximeter (defined as SpO2 < 92%) [13], the intubation attempt will be stopped and the lungs will be ventilated with an oxygen-volatile anesthetic mixture for 3 min. A second attempt will be allowed with the randomly allocated airway device. If intubation is unsuccessful after two attempts, the protocol allows intubating the patient with the anesthesiologist's instrument of choice. [14]

The anesthesiologist will be asked to rate the ease of intubation using a 10 cm visual analog scale (0 for much of ease and 10 for extremely difficult). Hemodynamic parameters (heart rate, systolic and mean blood pressures) will be recorded at baseline, during the intubation process, and each 1-min for 5 min and 10 min after tracheal intubation.

A careful examination of the oropharynx will be performed after intubation to determine any lip, dental or mucosal trauma. Following recovery from anesthesia in the post-anesthesia care unit, a trained anesthesiologist who will not be involved in the study and who is blind to the device used will evaluate all patients for a postoperative sore throat to ensure consistency and severity.

Statistical Analysis

Data will be tested for normality using the Kolmogorov-Smirnov test. Serial changes in the studied data at intubation will be analyzed with repeated-measures analysis of variance. Categorical data will be analyzed using Fischer's exact test. Repeated measure analysis of variance (ANOVA) will be used for continuous parametric variables and the differences will be then corrected by post-hoc Bonferoni test. The Kruskal-Wallis one-way ANOVA will be performed for intergroup comparisons for the non-parametric values and post hoc pairwise comparisons will be done using the Wilcoxon rank sum t test. p value < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status class I-II
* aged 18-65 years
* scheduled for elective surgery
* under general anesthesia

Exclusion Criteria:

* Expected or known difficult airway
* history of cervical spine injury
* history of cervical spine surgery
* previous throat surgery
* previous oral surgery
* gastro-esophageal reflux disease
* pregnancy
* need for rapid sequence induction
* emergent surgery
* body mass index higher than 35 kg/m2
* Missing incisor teeth
* Unstable hypertension
* Unstable coronary artery disease
* Asthma
* Cerbrovascular disease

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2013-09; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Time to tracheal intubation | participants will be followed for the duration of tracheal intubation, an expected average of 60 seconds
  the time when the investigated laryngoscope passes the central incisors to the time when the tip of the tracheal tube passed through the glottis

SECONDARY OUTCOMES:
laryngoscopic view | participants will be followed for the duration of laryngeal exposure, an expected average of 90 seconds
  The best view during laryngoscopy (using Cormack and Lehane classification)
ease of intubation | participants will be followed for the duration of tracheal intubation, an expected average of 60 seconds
  using a 10 cm visual analog scale (0 for much of ease and 10 for extremely difficult).
number of intubation attempts | participants will be followed for the duration of tracheal intubation, an expected average of 60 seconds
  number of intubation attempts
number of optimization maneuvers | participants will be followed for the duration of tracheal intubation, an expected average of 60 seconds
  If intubation is unsuccessful at the first attempt, took longer than 120 seconds, or if desaturation noted on the pulse oximeter (defined as SpO2 < 92%) [14], the intubation attempt will be stopped and the lungs will be ventilated with an oxygen-volatile anesthetic mixture for 3 min. A second attempt will be allowed with the randomly allocated airway device.
duration of laryngoscopy | during laryngoscopy
  the time from holding of the investigated laryngoscope to the appearance of as the first upward deflection on the capnograph
Hemodynamic parameters | participants will be followed for the duration of laryngeal exposure, an expected average of 90 seconds
  heart rate, systolic and mean blood pressures

CONTACTS AND LOCATIONS:
Overall Officials: Abdulmohsen Al Ghamdi, MD, Principal Investigator — Associate Professor/Chairman of Anesthesiology; Mohamed R El Tahan, MD, Study Director — Associate Professor of Anesthesiology; Alaa M Khidr, MD, Study Chair — Assistant Professor of Anesthesiology
Locations (2):
- Saudi Arabia (2):
  - Dammam University, Khobar, Eastern Province
  - King Fahd Hospital of the University, Khobar, Eastern Province